CLINICAL TRIAL: NCT03555357
Title: Platelet Rich Therapy for Scar Revision Post Abdominoplasty
Brief Title: Platelet Rich Therapy for Scar Revision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rejuva Medical Aesthetics (Other)
Responsible Party: Principal Investigator, Alex Reivitis, Clinical Research Coordinator, Rejuva Medical Aesthetics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF02
Record Dates: First submitted 2018-05-08; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Abdominoplasty Scar Revision
Keywords: Abdomen; Abdominoplasty; Scar Therapy; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: Subjects will receive both PRP and PRF injections to the scar. One side will be assigned to PRP and the other PRF (randomly assigned by Clinical Research Coordinator).
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will not be aware of which side is treated with PRP vs. PRF. The blind observer will also not be informed which side was treated with PRP vs. PRF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Active Comparator): Platelet Rich Plasma (PRP) injections into one half of the scar will be preformed. PRP is already considered an effective treatment for scar therapy.This will be randomly assigned by the clinical research coordinator .
  Interventions: Other: Platelet Rich Plasma
- PRF (Experimental): Platelet Rich Fibrin (PRF) injections will be preformed the other half of the scar that is not treated with PRP. PRF has not been established as an effective scar treatment. The PRF will be considered experimental as this study seeks to evaluate if it is more effective than PRP.
  Interventions: Other: Platelet Rich Fibrin

INTERVENTIONS:
Other: Platelet Rich Fibrin — Platelet Rich Fibrin (PRF) is the next generation of PRP and contains very high concentrations white blood cells, fibrin and a small amount of mesenchymal stem cells found circulating in our bloodstreams. Due to a lack of anticoagulant in the tube, PRF becomes a gel after 15-20 minutes of being isolated. These properties make PRF useful in reconstructive and aesthetic medicine but may also be beneficial for scar therapy in the same way PRP is currently used.
  Other Names: PRF
  Arms: PRF
Other: Platelet Rich Plasma — Platelet Rich Plasma (PRP) has been used in surgical settings to stimulate healing and promote tissue regeneration. In the field of cosmetic medicine, PRP has been used topically or as an injection to stimulate collagen production and enhance the efficacy of cosmetic procedures such as fat transfer, hair loss therapies, laser treatments, and microneedling. Harvested PRP has platelets, fibrin, and white blood cells, which contribute to wound healing, neocollagenesis, and elastogenesis
  Other Names: PRP
  Arms: PRP

SUMMARY:
This study will evaluate the efficacy of platelet injections for use of scar therapy post abdominoplasty operations.

DETAILED DESCRIPTION:
Platelet therapy is quickly becoming an integral aspect of both medical and cosmetic procedures. Most notably, Platelet Rich Plasma (PRP) has been used in surgical settings to stimulate healing and promote tissue regeneration. In the field of cosmetic medicine, PRP has been used topically or as an injection to stimulate collagen production and enhance the efficacy of cosmetic procedures such as fat transfer, hair loss therapies, laser treatments, and microneedling. Harvested PRP has platelets, fibrin, and white blood cells, which contribute to wound healing, neocollagenesis, and elastogenesis. Platelet Rich Fibrin (PRF) is the next generation of PRP and contains very high concentrations white blood cells, fibrin and a small amount of mesenchymal stem cells found circulating in our bloodstreams. Due to a lack of anticoagulant in the tube, PRF becomes a gel after 15-20 minutes of being isolated. These properties make PRF useful in reconstructive and aesthetic medicine but may also be beneficial for scar therapy in the same way PRP is currently used.The purpose of this study is to evaluate the efficacy of platelet rich plasma vs. platelet rich fibrin for scar therapy in abdominoplasty who are at least one-year post operation.

ELIGIBILITY:
Inclusion Criteria:

* Ten (10) subjects
* male and female abdominoplasty procedures at least one year ago.
* must be able to provide healthy blood sample
* must be available for the duration of the study and all follow ups (12 months).

Exclusion Criteria:

* Pregnant and breast-feeding patients are not eligible for this study due to unstudied effects of injectables on the growing fetus and/or breast milk.
* patients who have undergone other scar therapies for the same scar.
* chronic health problems that may prevent the investigators from obtaining a viable blood sample,
* topical infection,
* any subjects who intend to have other scar procedures during the timeline of the study (12 months including punch biopsy procedures 3 months post treatment and 6 months post treatment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetics Improvement Scale (GAIS) | 6 months
  Blind observer will complete the Global Aesthetics Improvement Scale at 6 months. The scale is from 1-5, where 1 is greatly improved cosmetic outcome and 5 is worsened cosmetic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kian Karimi, MD,FACS, Principal Investigator — Rejuva Medical Aesthetics

IPD SHARING:
Plan to Share IPD: No